CLINICAL TRIAL: NCT02638948
Title: Phase 2, Randomized, Multi-Center, Double-Blind, Dose-Ranging, Placebo Controlled, Adaptive Design Study to Evaluate the Efficacy and Safety/Pharmacokinetics of BMS-986142 in Subjects With Moderate to Severe Rheumatoid Arthritis With an Inadequate Response to Methotrexate With or Without TNF Inhibitors
Brief Title: Efficacy and Safety Study of BMS-986142 in Patients With Moderate to Severe Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM006-016; 2015-002887-17 (EudraCT Number)
Record Dates: First submitted 2015-12-21; First posted 2015-12-23 (Estimated); Results first posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo + Methotrexate dose as specified
  Interventions: Drug: Placebo; Drug: Methotrexate
- Dose Level 1 (Experimental): BMS-986142 at dose level 1+ Methotrexate as specified
  Interventions: Drug: BMS-986142; Drug: Methotrexate
- Dose Level 2 (Experimental): BMS-986142 at dose level 2 + Methotrexate as specified
  Interventions: Drug: BMS-986142; Drug: Methotrexate

INTERVENTIONS:
Drug: BMS-986142 — BMS986142 specific dose on specific days
  Arms: Dose Level 1; Dose Level 2
Drug: Placebo — Placebo of BMS-986142 specific dose on specific days
  Arms: Placebo
Drug: Methotrexate — Methotrexate specific dose on specific days

SUMMARY:
The purpose of this study is to determine whether the study drug, BMS-986142, is safe and effective in treating moderate to severe rheumatoid arthritis in subjects with an inadequate response to methotrexate or methotrexate and up to 2 tumour necrosis factor (TNF) Inhibitors. Patients who qualify will be randomized to either one of 3 doses of BMS-986142 or placebo in 1:1:1 randomization for 12 weeks. Disease activity and safety will be assessed over the course of the study.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Male and female age 18 and above
* Diagnosed with active rheumatoid arthritis (RA) by standard criteria at least 16 weeks before screening, have functional ACR class I-III
* Have an inadequate response to methotrexate
* In addition to an inadequate response to methotrexate have an inadequate response or intolerance to 1 but not more than 2 TNF inhibitors
* Have a minimum of 6 swollen and 6 tender joints (from 66/68 joint count)
* Have hsCRP of ≥ 0.8 mg/dL (8mg/L) [by central laboratory values] or an ESR ≥ 28 mm/hr
* Willing to use effective birth control for the entire length of the study

Exclusion Criteria:

* Diagnosed with juvenile Rheumatoid Arthritis
* Have been treated with other biologic treatment than a TNF inhibitor
* Active systemic bacterial, viral or fungal infection or evidence of prior or current Hepatitis B or C infection or HIV infection, latent bacterial, viral or fungal infections
* Have been treated with Intramuscular or Intra-articular glucocorticosteroids within 4 weeks of randomization
* Taking Oral steroids at dose above 10 mg/day of prednisone (or prednisone equivalents)
* Have other autoimmune disease other than RA like lupus, multiple sclerosis
* Have significant concurrent medical condition at the time of screening or baseline visit

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (97):
- United States (26):
  - Rheumatology Associates Of North Alabama, P.C., Huntsville, Alabama
  - St. Joseph Heritage Medical Group, Fullerton, California
  - C.V Mehta M.D Medical Corp, Hemet, California
  - HCP Clinical Research, LLC, Huntington Beach, California
  - Leon Medical Research, Miami, Florida
  - San Marcus Research Clinic, Inc., Miami, Florida
  - Coral Research Clinic Corp, Miami, Florida
  - Precision Research Organization, Miami Lakes, Florida
  - The Arthritis Center, Palm Harbor, Florida
  - Vizae Clinical Trials Management, Pembroke Pines, Florida
  - Integral Rheumatology & Immunology Specialists, Plantation, Florida
  - North Georgia Rheumatology Group, Lawrenceville, Georgia
  - Arthritis And Diabetes Clinic, Monroe, Louisiana
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Aa Mrc Llc, Grand Blanc, Michigan
  - Albuquerque Center For Rheumatology, Albuquerque, New Mexico
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Paramount Medical Research & Consulting, Llc, Middleburg Heights, Ohio
  - East Penn Rheumatology, Bethlehem, Pennsylvania
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Advanced Rheumatology & Arthritis Research Center, P.C, Wexford, Pennsylvania
  - Local Institution, Wyomissing, Pennsylvania
  - West Tennessee Research Institute, Jackson, Tennessee
  - Pharma Tex Research, Amarillo, Texas
  - Tekton Research Inc, Austin, Texas
  - Southwest Rheumatology Research LLC, Mesquite, Texas
- Argentina (4):
  - Local Institution, Capital Federal, Buenos Aires
  - Aprillus Asistencia e Investigacion, Capital Federal, Buenos Aires
  - Instituto De Rehabilitacion Psicofisica, Buenos Aires
  - Instituto Reumatologico Strusberg, Córdoba
- Universitaetsklinik Fuer Innere Medizin 3, Vienna, Austria
- Brazil (6):
  - Local Institution, Goiânia, Goiás
  - Local Institution, Juiz de Fora, Minas Gerais
  - Local Institution, Curitiba, Paraná
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Santo André, São Paulo
  - Local Institution, São Paulo
- Canada (2):
  - Aggarwal And Associates, Brampton, Ontario
  - Dr. Anil K Gupta Med Prof Corp, Toronto, Ontario
- France (4):
  - Local Institution, Corbeil-Essonnes
  - Local Institution, Montpellier
  - Local Institution, Orléans
  - Local Institution, Strasbourg
- Germany (3):
  - Asklepios Gesundheitszentrum, Elmshorn
  - Medizinsche Universitaetsklinik Freiburg, Freiburg im Breisgau
  - Smo.Md Gmbh, Magdeburg
- Italy (2):
  - Local Institution, Florence
  - Local Institution, Padua
- Japan (19):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Fukuoka, Fukuoka
  - Local Institution, Kitakyushu-shi, Fukuoka
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Kato-shi, Hyōgo
  - Local Institution, Sagamihara-shi, Kanagawa
  - Local Institution, Kumamoto, Kumamoto
  - Local Institution, Sendai, Miyagi
  - Local Institution, Sasebo-shi, Nagasaki
  - Local Institution, Kawachi-Nagano, Osaka
  - Local Institution, Osaka, Osaka
  - Local Institution, Iruma-gun, Saitama
  - Local Institution, Kawagoe-shi, Saitama
  - Local Institution, Hamamatsu, Shizuoka
  - Local Institution, Chuo-ku, Tokyo
  - Local Institution, Itabashi-ku, Tokyo
  - Local Institution, Meguro-ku, Tokyo
  - Local Institution, Shinjuku-Ku, Tokyo
  - Local Institution, Osaki-shi
- Mexico (7):
  - CINTRE - Centro de investigacion y tratamiento reumatologico, S.C., Mexico City, Distrito Fededral
  - Consultorio Privado de Especialidad, Guadalajara, Jalisco
  - Clinica de Investigacion en Reumatologia y Obesidad S.C., Guadalajara, Jalisco
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Villahermosa, Tabasco
  - Unidad Reumatologica Las Americas, S.C. P., Mérida, Yucatán
  - Centro de Alta Especialidad en Reumatologia e Investigacion del Potosi S.C., Distrito Federal
- Maasstad Ziekenhuis Rotterdam, Rotterdam, Netherlands
- Poland (8):
  - Nzoz Osteo-Medic S.C. A. Racewicz, J.Supronik, Bialystok
  - Local Institution, Bialystok
  - Centrum Badan Klinicznych JCI Life Science Park, Krakow
  - Local Institution, Lublin
  - Local Institution, Nadarzyn
  - Local Institution, Poznan
  - Local Institution, Warsaw
  - Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji, Warsaw
- Russia (3):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
  - Local Institution, Tolyatti
- South Africa (4):
  - Local Institution, Benoni, Gauteng
  - Local Institution, Cape Town, Western Cape
  - Local Institution, George, Western Cape
  - Local Institution, Somerset West, Western Cape
- South Korea (2):
  - Local Institution, Daegu
  - Local Institution, Seoul
- Spain (3):
  - Local Institution, A Coruña
  - Fundacion Jimenez Diaz, Madrid
  - Local Institution, Santiago Compostela
- Taiwan (2):
  - Local Institution, Taichung
  - Local Institution, Taipei

REFERENCES:
- [Derived] Conaghan PG, Nowak M, Du S, Luo Y, Landis J, Pachai C, Fura A, Catlett IM, Grasela DM, Ostergaard M. Evaluation of BMS-986142, a reversible Bruton's tyrosine kinase inhibitor, for the treatment of rheumatoid arthritis: a phase 2, randomised, double-blind, dose-ranging, placebo-controlled, adaptive design study. Lancet Rheumatol. 2023 May;5(5):e263-e273. doi: 10.1016/S2665-9913(23)00089-9. PMID 38251590
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 508 participants who signed the informed consent form and were enrolled in the study; 248 participants were randomized, and 247 participants were administered study drug (1 participant did not take any double-blind study medication).
Groups:
- Placebo: Oral dose of matching placebo for BMS-986142 was administered daily for 12 weeks.
- BMS 100mg: Oral dose of BMS-986142 100mg was administered daily for 12 weeks.
- BMS 200mg: Oral dose of BMS-986142 200mg was administered daily for 12 weeks.
- BMS 350mg: Oral dose of BMS-986142 350mg was administered daily for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | BMS 100mg | BMS 200mg | BMS 350mg
Started | 75 | 73 | 73 | 26
Completed | 66 | 62 | 66 | 18
Not Completed | 9 | 11 | 7 | 8
Not completed — Withdrawal by Subject | 4 | 5 | 3 | 1
Not completed — Administrative Reason by Sponsor | 0 | 1 | 0 | 4
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Lack of Efficacy | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1
Not completed — Poor/Non-Compliance | 0 | 2 | 1 | 0
Not completed — Participant no longer met study criteria | 0 | 1 | 0 | 0
Not completed — Other than specified above | 4 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized and treated participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BMS 100mg | BMS 200mg | BMS 350mg | Total
Number analyzed (Participants) | 75 | 73 | 73 | 26 | 247
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.6 (11.61) | 57.6 (13.01) | 55.2 (13.13) | 52.9 (13.16) | 56.7 (12.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 67 | 62 | 21 | 214
  Male | 11 | 6 | 11 | 5 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 24 | 28 | 10 | 84
  Not Hispanic or Latino | 27 | 24 | 25 | 8 | 84
  Unknown or Not Reported | 26 | 25 | 20 | 8 | 79
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 52 | 54 | 58 | 24 | 188
  Black or African American | 6 | 9 | 5 | 1 | 21
  Asian | 14 | 8 | 8 | 1 | 31
  Other | 3 | 2 | 2 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response at Week 12
Description: ACR responses are assessed with a composite rating scale of the American College of Rheumatology that includes 7 variables: tender joint count (TJC); swollen joint count (SJC); levels of an acute phase reactant C-reactive Protein levels (CRP); participant's assessment of pain; participant's global assessment of disease activity; physician's global assessment of disease activity; participant's assessment of physical function by health assessment questionnaire disability index (HAQ-DI). ACR20 is defined as achieving at least 20% improvement in both TJC and SJC, and at least 20% improvement in at least 3 of the 5 other assessments of the ACR. Percentage of Participants achieving ACR20 = (number of participants with measure/event of interest)/(number of particpants in the analysis)*100
Time Frame: Week 12
Population: Analysis was performed on efficacy population which excluded participants who were randomized to a treatment arm and discontinued based on the interim analysis (IA).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | BMS 100mg | BMS 200mg | BMS 350mg
Number analyzed (Participants) | 75 | 73 | 73 | 26
Percentage of participants | 30.7 [20.2 to 41.1] | 35.6 [24.6 to 46.6] | 42.5 [31.1 to 53.8] | 30.8 [13.0 to 48.5]
Statistical Analysis 1: Comparison: Placebo vs BMS 100mg; Test type: Superiority; p = 0.5224, Chi-squared — Threshold for significance = 0.05; Estimate of Difference (%) = 4.9, 95% CI 2-sided [-10.2 to 20.1]
Statistical Analysis 2: Comparison: Placebo vs BMS 200mg; Test type: Superiority; p = 0.1360, Chi-squared — Threshold for significance = 0.05; Estimate of Difference (%) = 11.8, 95% CI 2-sided [-3.6 to 27.2]
Statistical Analysis 3: Comparison: Placebo vs BMS 350mg; Test type: Superiority; p = 0.9922, Chi-squared — Threshold for significance = 0.05; Estimate of Difference (%) = 0.1, 95% CI 2-sided [-20.5 to 20.7]

2. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response at Week 12
Description: ACR responses are assessed with a composite rating scale of the American College of Rheumatology that includes 7 variables: TJC; SJC; levels of an acute phase reactant (CRP level); participant's assessment of pain; participant's global assessment of disease activity; physician's global assessment of disease activity; participant's assessment of physical function by HAQ--DI. ACR70 is defined as achieving at least 70% improvement in both TJC and SJC, and at least 70% improvement in at least 3 of the 5 other assessments of the ACR. Percentage of Participants achieving ACR70 = (number of participants with measure/event of interest)/(number of particpants in the analysis)*100
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | BMS 100mg | BMS 200mg | BMS 350mg
Number analyzed (Participants) | 75 | 73 | 73 | 26
Percentage of participants | 4.0 [0.8 to 11.2] | 4.1 [0.9 to 11.5] | 9.6 [2.8 to 16.3] | 3.8 [0.1 to 19.6]
Statistical Analysis 1: Comparison: Placebo vs BMS 100mg; Test type: Superiority; p = 1.0000, Chi-squared — Threshold for significance = 0.05; Estimate of Difference (%) = 0.1, 95% CI 2-sided [-16.0 to 16.5]
Statistical Analysis 2: Comparison: Placebo vs BMS 200mg; Test type: Superiority; p = 0.2058, Chi-squared — Threshold for significance = 0.05; Estimate of Difference (%) = 5.6, 95% CI 2-sided [-10.5 to 21.9]
Statistical Analysis 3: Comparison: Placebo vs BMS 350mg; Test type: Superiority; p = 1.0000, Chi-squared — Threshold for significance = 0.05; Estimate of Difference (%) = -0.2, 95% CI 2-sided [-22.5 to 22.2]

3. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% Response Over Time From Baseline to Week 12
Description: as for outcome 1
Time Frame: Baseline, Day 15, Day 29, Day 57, Day 85
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | BMS 100mg | BMS 200mg | BMS 350mg
Number analyzed (Participants) | 75 | 73 | 73 | 26
Percentage of participants
  Baseline (Day 1) | 0.0 [NA to NA] — Here 'NA' signifies not estimable (NE): number of participants with ACR20% response was zero due to which 95% confidence interval was NE | 0.0 [NA to NA] — Here 'NA' signifies not estimable (NE): number of participants with ACR20% response was zero due to which 95% confidence interval was NE | 0.0 [NA to NA] — Here 'NA' signifies not estimable (NE): number of participants with ACR20% response was zero due to which 95% confidence interval was NE | 0.0 [NA to NA] — Here 'NA' signifies not estimable (NE): number of participants with ACR20% response was zero due to which 95% confidence interval was NE
  Day 15 | 10.7 [3.7 to 17.7] | 13.7 [5.8 to 21.6] | 24.7 [14.8 to 34.5] | 15.4 [4.4 to 34.9]
  Day 29 | 18.7 [9.8 to 27.5] | 23.3 [13.6 to 33.0] | 21.9 [12.4 to 31.4] | 26.9 [9.9 to 44.0]
  Day 57 | 28.0 [17.8 to 38.2] | 41.1 [29.8 to 52.4] | 39.7 [28.5 to 51.0] | 15.4 [4.4 to 34.9]
  Day 85 | 30.7 [20.2 to 41.1] | 35.6 [24.6 to 46.6] | 42.5 [31.1 to 53.8] | 30.8 [13.0 to 48.5]

4. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response Over Time From Baseline to Week 12
Description: ACR responses are assessed with a composite rating scale of the American College of Rheumatology that includes 7 variables: TJC; SJC; levels of an acute phase reactant (CRP level); participant's assessment of pain; participant's global assessment of disease activity; physician's global assessment of disease activity; participant's assessment of physical function by HAQ--DI. ACR70 is defined as achieving at least 50% improvement in both TJC and SJC, and at least 50% improvement in at least 3 of the 5 other assessments of the ACR. Percentage of Participants achieving ACR50 = (number of participants with measure/event of interest)/(number of particpants in the analysis)*100
Time Frame: Baseline, Day 15, Day 29, Day 57, Day 85
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | BMS 100mg | BMS 200mg | BMS 350mg
Number analyzed (Participants) | 75 | 73 | 73 | 26
Percentage of participants
  Baseline (Day 1) | 0 [NA to NA] — Here 'NA' signifies not estimable (NE): number of participants with ACR50% response was zero due to which 95% confidence interval was NE | 0 [NA to NA] — Here 'NA' signifies not estimable (NE): number of participants with ACR50% response was zero due to which 95% confidence interval was NE | 0 [NA to NA] — Here 'NA' signifies not estimable (NE): number of participants with ACR50% response was zero due to which 95% confidence interval was NE | 0 [NA to NA] — Here 'NA' signifies not estimable (NE): number of participants with ACR50% response was zero due to which 95% confidence interval was NE
  Day 15 | 2.7 [0.3 to 9.3] | 4.1 [0.9 to 11.5] | 5.5 [1.5 to 13.4] | 3.8 [0.1 to 19.6]
  Day 29 | 2.7 [0.3 to 9.3] | 4.1 [0.9 to 11.5] | 6.8 [1.1 to 12.6] | 7.7 [0.9 to 25.1]
  Day 57 | 9.3 [2.7 to 15.9] | 12.3 [4.8 to 19.9] | 13.7 [5.8 to 21.6] | 7.7 [0.9 to 25.1]
  Day 85 | 9.3 [2.7 to 15.9] | 13.7 [5.8 to 21.6] | 16.4 [7.9 to 24.9] | 11.5 [2.4 to 30.2]

5. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% Response Over Time From Baseline to Week 12
Description: as for outcome 2
Time Frame: Baseline, Day 15, Day 29, Day 57, Day 85
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | BMS 100mg | BMS 200mg | BMS 350mg
Number analyzed (Participants) | 75 | 73 | 73 | 26
Percentage of participants
  Baseline (Day 1) | 0 [NA to NA] — Here 'NA' signifies not estimable (NE): number of participants with ACR70% response was zero due to which 95% confidence interval was NE | 0 [NA to NA] — Here 'NA' signifies not estimable (NE): number of participants with ACR70% response was zero due to which 95% confidence interval was NE | 0 [NA to NA] — Here 'NA' signifies not estimable (NE): number of participants with ACR70% response was zero due to which 95% confidence interval was NE | 0 [NA to NA] — Here 'NA' signifies not estimable (NE): number of participants with ACR70% response was zero due to which 95% confidence interval was NE
  Day 15 | 1.3 [0.0 to 7.2] | 0.0 [0.0 to 4.9] | 1.4 [0.0 to 7.4] | 0.0 [0.0 to 13.2]
  Day 29 | 0.0 [NA to NA] — Here 'NA' signifies not estimable (NE): number of participants with ACR70% response was zero due to which 95% confidence interval was NE. | 0.0 [NA to NA] — Here 'NA' signifies NE: number of participants with ACR70% response was zero due to which 95% confidence interval was NE. | 0.0 [NA to NA] — Here 'NA' signifies NE: number of participants with ACR70% response was zero due to which 95% confidence interval was NE. | 0.0 [NA to NA] — Here 'NA' signifies NE: number of participants with ACR70% response was zero due to which 95% confidence interval was NE.
  Day 57 | 1.3 [0.0 to 7.2] | 5.5 [1.5 to 13.4] | 5.5 [1.5 to 13.4] | 3.8 [0.1 to 19.6]
  Day 85 | 4.0 [0.8 to 11.2] | 4.1 [0.9 to 11.5] | 9.6 [2.8 to 16.3] | 3.8 [0.1 to 19.6]

6. Secondary Outcome: Percentage of Participants Achieving < 2.6 Response in Disease Activity Score for 28 Joints -C-Reactive Protein (DAS28--CRP) Score at Week 12
Description: DAS28 is a composite score that includes 4 variables: TJC (based on 28 joints); SJC (based on 28 joints); General health (GH) assessment by the participant assessed from the ACR rheumatoid arthritis (RA) core set questionnaire (participant global assessment) in 100 mm visual analog scale (VAS). Marker of inflammation assessed by the high sensitivity C-reactive protein (hs-CRP) in mg/L. The DAS28 score provides a number indicating the current disease activity of the RA. DAS28 total score ranges from 2-10. A DAS28 score above 5.1 means high disease activity, whereas a DAS28 score below 3.2 indicates low disease activity and a DAS28 score below 2.6 means disease remission.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | BMS 100mg | BMS 200mg | BMS 350mg
Number analyzed (Participants) | 75 | 73 | 73 | 26
Percentage of participants | 6.7 [1.0 to 12.3] | 9.6 [2.8 to 16.3] | 11.0 [3.8 to 18.1] | 0.0 [0.0 to 13.2]

7. Secondary Outcome: Percentage of Participants Achieving < 2.6 Response in Disease Activity Score for 28 Joints Erythrocyte Sedimentation Rate (DAS28--ESR) Score at Week 12
Description: DAS28-ESR is a composite score that includes 4 variables: TJC (based on 28 joints); SJC (based on 28 joints); General health (GH) assessment by the participant assessed from the ACR RA core set questionnaire (participant global assessment) in 100 mm VAS; Marker of inflammation assessed by ESR in mm/hr. The DAS28-ESR score provides a number indicating the current disease activity of the RA. DAS28-ESR total score ranges from 2-10. A DAS28-ESR score above 5.1 means high disease activity, DAS28-ESR score below 3.2 indicates low disease activity and DAS28-ESR score below 2.6 means disease remission.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | BMS 100mg | BMS 200mg | BMS 350mg
Number analyzed (Participants) | 75 | 73 | 73 | 26
Percentage of participants | 0.0 [0.0 to 4.8] | 6.8 [1.1 to 12.6] | 1.4 [0.0 to 7.4] | 0.0 [0.0 to 13.2]

8. Secondary Outcome: Percentage of Participants Achieving <= 2.8 Response in Clinical Disease Activity Index (CDAI) Score at Week 12
Description: CDAI is a composite index constructed to measure clinical remission in RA that does not include a laboratory test, and is a numerical summation of 4 components: TJC (28 joints), SJC (28 joints), Participant's Global Assessment of Disease Activity VAS (in cm), and Physician's Global Assessment of Disease VAS (in cm). Total scores ranges from 0 to 76 with a negative change in CDAI score indicating an improvement in disease activity and a positive change in score indicating a worsening of disease activity.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | BMS 100mg | BMS 200mg | BMS 350mg
Number analyzed (Participants) | 75 | 73 | 73 | 26
Percentage of participants | 0.0 [0.0 to 4.8] | 6.8 [1.1 to 12.6] | 6.8 [1.1 to 12.6] | 0.0 [0.0 to 13.2]

9. Secondary Outcome: Percentage of Participants Achieving <= 3.3 Response in Simple Disease Activity Index (SDAI) Score at Week 12
Description: The SDAI is the numerical sum of five outcome parameters: TJC and SJC based on a 28-joint assessment, patient global assessment (PtGA) and physician global assessment (PGA) assessed on a VAS scale ranging from 0 to 10 cm, where higher scores indicate greater affection due to disease activity, and CRP measured in terms of milligram per deciliter (mg/dL). SDAI total score ranges from 0 to 86. SDAI <= 3.3 indicates disease remission, > 3.4 to 11 indicates low disease activity, >11 to 26 indicates moderate disease activity, and >26 indicates high disease activity.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | BMS 100mg | BMS 200mg | BMS 350mg
Number analyzed (Participants) | 75 | 73 | 73 | 26
Percentage of participants | 0.0 [0.0 to 4.8] | 6.8 [1.1 to 12.6] | 6.8 [1.1 to 12.6] | 0.0 [0.0 to 13.2]

10. Secondary Outcome: Percentage of Participants Achieving Boolean Remission Criteria at Week 12
Description: Boolean remission criteria was defined as: tender joint count28 <= 1; swollen joint count28 <= 1; physician's global assessment <= 1; and CRP <= 1 mg/deciliter.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | BMS 100mg | BMS 200mg | BMS 350mg
Number analyzed (Participants) | 75 | 73 | 73 | 26
Percentage of participants | 1.3 [0.0 to 7.2] | 4.1 [0.9 to 11.5] | 4.1 [0.9 to 11.5] | 0.0 [0.0 to 13.2]

11. Secondary Outcome: Change From Baseline in DAS28-CRP Score Over Time up to Week 12
Description: as for outcome 6
Time Frame: Baseline, Day 85 (Week 12)
Population: Analysis was performed on efficacy population which excluded participants who were randomized to a treatment arm and discontinued based on the interim analysis (IA). Here 'N' signifies number of participants analyzed who were evaluable for this outcome measure.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | BMS 100mg | BMS 200mg | BMS 350mg
Number analyzed (Participants) | 64 | 63 | 64 | 15
Units on a scale | -1.1 (0.141) | -1.1 (0.176) | -1.4 (0.168) | -1.4 (0.194)

12. Secondary Outcome: Change From Baseline in DAS28-ESR Score Over Time up to Week 12
Description: as for outcome 7
Time Frame: Baseline, Week 12
Population: as for outcome 11
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | BMS 100mg | BMS 200mg | BMS 350mg
Number analyzed (Participants) | 64 | 63 | 65 | 14
Units on a scale | -1.1 (0.149) | -1.1 (0.166) | -1.4 (0.161) | -1.5 (0.247)

13. Secondary Outcome: Change From Baseline in CDAI Score Over Time up to Week 12
Description: as for outcome 8
Time Frame: Baseline, Week 12
Population: as for outcome 11
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | BMS 100mg | BMS 200mg | BMS 350mg
Number analyzed (Participants) | 65 | 61 | 68 | 16
Units on a scale | -14.9 (1.591) | -13.6 (2.030) | -16.0 (1.828) | -17.6 (2.519)

14. Secondary Outcome: Change From Baseline in SDAI Score Over Time up to Week 12
Description: The SDAI is the numerical sum of five outcome parameters: TJC and SJC based on a 28-joint assessment, PtGA and PGA assessed on a VAS scale ranging from 0 to 10 cm, where higher scores indicate greater affection due to disease activity, and CRP measured in terms of mg/dL. SDAI total score ranges from 0 to 86. SDAI <= 3.3 indicates disease remission, > 3.4 to 11 indicates low disease activity, >11 to 26 indicates moderate disease activity, and >26 indicates high disease activity.
Time Frame: Baseline, Week 12
Population: as for outcome 11
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | BMS 100mg | BMS 200mg | BMS 350mg
Number analyzed (Participants) | 64 | 61 | 64 | 15
Units on a scale | -14.8 (1.628) | -13.9 (2.090) | -16.6 (1.954) | -18.9 (3.218)

15. Secondary Outcome: Number of Participants With Adverse Events (AEs), and Serious AEs (SAEs)
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), persistent or significant disability/incapacity, or a congenital anomaly, or a medically important event.
Time Frame: Up to 30 days after treatment discontinuation
Population: All treated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BMS 100mg | BMS 200mg | BMS 350mg
Number analyzed (Participants) | 75 | 73 | 73 | 26
Participants
  AEs | 36 | 39 | 39 | 19
  SAEs | 4 | 2 | 0 | 0

16. Secondary Outcome: Trough Observed Plasma Concentration (Ctrough) of BMS-986142
Description: Ctrough was defined as trough observed plasma concentration.
Time Frame: Week 4, 8, and 12
Population: Analysis was performed on pharmacokinetic population which included all participants who received BMS-986142 and had any available concentration-time data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/mL
Arm/Group | BMS 100mg | BMS 200mg | BMS 350mg
Number analyzed (Participants) | 73 | 73 | 26
nanogram/mL
  Week 4: number analyzed (Participants) | 60 | 61 | 16
  Week 4 | 47.9 (119.0) | 111.8 (101.7) | 195.9 (91.9)
  Week 8: number analyzed (Participants) | 54 | 60 | 18
  Week 8 | 41.2 (95.3) | 92.2 (124.5) | 283.0 (133.3)
  Week 12: number analyzed (Participants) | 55 | 52 | 13
  Week 12 | 28.4 (123.0) | 75.6 (155.4) | 169.5 (83.2)

17. Secondary Outcome: Mean Change From Baseline in Rheumatoid Arthritis Magnetic Resonance Imaging Scoring System (RAMRIS) Scores for Synovitis at Week 4 and 12
Description: Synovitis is assessed in 3 wrist regions (A. the distal radioulnar joint; B. the radiocarpal joint; C. the intercarpal and carpometacarpophalangeal, CMC, joints) and in each MCP joint. For each wrist region, possible score ranges from 0-3, with 0=normal, 1=mild, 2=moderate, and 3=severe damage. The total synovitis score per wrist=the sum of the individual scores for the 3 wrist regions. Minimum score per wrist ranges from 0, indicating no damage, to 9 (score of 3*3 wrist regions), indicating most severe damage. A negative change from baseline indicates improvement.
Time Frame: Week 4 and Week 12
Population: Analysis was performed on efficacy population which excluded participants who were randomized to a treatment arm and discontinued based on the interim analysis (IA). Here number analyzed = number of randomized and treated participants with non-missing value at each time point
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | BMS 100mg | BMS 200mg | BMS 350mg
Number analyzed (Participants) | 75 | 73 | 73 | 26
Scores on a scale
  Week 4: number analyzed (Participants) | 68 | 66 | 70 | 23
  Week 4 | 0.1 (0.226) | -0.2 (0.202) | 0.1 (0.182) | 0.1 (0.558)
  Week 12: number analyzed (Participants) | 68 | 66 | 70 | 23
  Week 12 | 0.7 (0.467) | -0.0 (0.315) | -0.3 (0.263) | 0.9 (1.163)

18. Secondary Outcome: Mean Change From Baseline in Rheumatoid Arthritis Magnetic Resonance Imaging Scoring System (RAMRIS) Scores for Osteitis at Week 4 and 12
Description: Osteitis was assessed at a total of 23 anatomic locations: 15 in 1 wrist and 8 in the hand of the same side. Each site is scored in 1.0 increments from 0 to 3, indicating involvement of original articular bone. The total score for the hands/wrists is the sum of the individual scores for each location. Thus the maximum score achievable per hand/wrist is 23 (total number of anatomic locations) * 3 (maximum per joint)=69. Minimum score=0, indicating normal. Increasing score=greater severity. A negative change from baseline indicates improvement.
Time Frame: Week 4, and Week 12
Population: as for outcome 17
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | BMS 100mg | BMS 200mg | BMS 350mg
Number analyzed (Participants) | 75 | 73 | 73 | 26
Scores on a scale
  Week 4: number analyzed (Participants) | 64 | 65 | 69 | 22
  Week 4 | 0.1 (0.223) | 0.2 (0.262) | 0.1 (0.148) | -0.1 (0.249)
  Week 12: number analyzed (Participants) | 64 | 65 | 69 | 22
  Week 12 | 0.4 (0.574) | 0.5 (0.451) | 0.0 (0.257) | 0.2 (0.654)

19. Secondary Outcome: Mean Change From Baseline in Rheumatoid Arthritis Magnetic Resonance Imaging Scoring System (RAMRIS) Scores for Bone Erosion at Week 4 and 12
Description: Bone erosion assessed at a total of 23 anatomic locations: 15 in 1 wrist and 8 in the hand of the same side. Each site is scored in 1.0 increments from 0 (no damage) to 10 (severe damage) according to erosion of the original articular bone (each unit=10% loss of articular bone). The total erosion score for the hands/wrists is the sum of the individual scores for each location. Thus the maximum score achievable per hand/wrist is 230. Increasing score=greater severity.A negative change from baseline indicates improvement.
Time Frame: Week 4 and Week 12
Population: as for outcome 17
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | BMS 100mg | BMS 200mg | BMS 350mg
Number analyzed (Participants) | 75 | 73 | 73 | 26
Scores on a scale
  Week 4: number analyzed (Participants) | 69 | 67 | 70 | 23
  Week 4 | 0.1 (0.048) | 0.1 (0.089) | -0.0 (0.036) | 0.0 (0.030)
  Week 12: number analyzed (Participants) | 69 | 67 | 70 | 23
  Week 12 | 0.1 (0.048) | 0.3 (0.248) | 0.0 (0.046) | 0.1 (0.072)

20. Secondary Outcome: Mean Change From Baseline in Rheumatoid Arthritis Magnetic Resonance Imaging Scoring System (RAMRIS) Scores for Cartilage Loss at Week 4 and 12
Description: Cartilage loss was assessed by MRI. Scans of 25 joints were read and scored for each participant by assessors. Scores for each location ranged 0-4 on a 9-point scale, with 0= no cartilage loss and 4= complete cartilage loss. Total score was the sum of the 25 individual scores and ranged 0-100 with 0= no cartilage loss and 100= most severe cartilage loss. A negative change from baseline indicates improvement.
Time Frame: Week 4, and Week12
Population: as for outcome 17
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | BMS 100mg | BMS 200mg | BMS 350mg
Number analyzed (Participants) | 75 | 73 | 73 | 26
Scores on a scale
  Week 4: number analyzed (Participants) | 69 | 67 | 70 | 23
  Week 4 | 0.1 (0.105) | 0.0 (0.064) | -0.0 (0.079) | 0.4 (0.169)
  Week 12: number analyzed (Participants) | 69 | 67 | 70 | 23
  Week 12 | 0.0 (0.116) | 0.3 (0.139) | 0.0 (0.111) | 0.5 (0.294)

ADVERSE EVENTS:
Time Frame: All Adverse Events were collected from signature of the informed consent until 30 days after last treatment administration. (Approximately 26 months)
Groups:
- BMS-986142 100mg: Oral dose of BMS-986142 100mg was administered daily for 12 weeks.
- BMS-986142 200mg: Oral dose of BMS-986142 200mg was administered daily for 12 weeks.
- BMS-986142 350mg: Oral dose of BMS-986142 350mg was administered daily for 12 weeks.
Arm/Group | BMS-986142 100mg | BMS-986142 200mg | BMS-986142 350mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/73 | 0/26 | 0/75
Serious Adverse Events (participants affected / at risk) | 2/73 | 0/73 | 0/26 | 4/75
Other Adverse Events (participants affected / at risk) | 12/73 | 17/73 | 14/26 | 11/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-986142 100mg (N=73) | BMS-986142 200mg (N=73) | BMS-986142 350mg (N=26) | Placebo (N=75)
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Open globe injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-986142 100mg (N=73) | BMS-986142 200mg (N=73) | BMS-986142 350mg (N=26) | Placebo (N=75)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 2 | 1
Nasopharyngitis (Infections and infestations) | 4 | 3 | 0 | 2
Urinary tract infection (Infections and infestations) | 5 | 6 | 5 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 5 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 2 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 4 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 3 | 6 | 2
Headache (Nervous system disorders) | 2 | 4 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period <=60 days from submitting for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2017-10-29): https://cdn.clinicaltrials.gov/large-docs/48/NCT02638948/Prot_000.pdf
  • Statistical Analysis Plan (2015-12-04): https://cdn.clinicaltrials.gov/large-docs/48/NCT02638948/SAP_001.pdf